CLINICAL TRIAL: NCT02463799
Title: A Phase 2 Study of Sipuleucel-T With or Without Radium-223 in Men With Asymptomatic or Minimally Symptomatic Bone-Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Study of Sipuleucel-T W/ or W/O Radium-223 in Men With Asymptomatic or Minimally Symptomatic Bone-MCRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Dendreon (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1522; IRB00056435 (Other: JHM IRB)
Record Dates: First submitted 2015-05-21; First posted 2015-06-04 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
Keywords: prostatic neoplasms; castration-resistant; bone metastasis; radium-223; sipuleucel-T
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radium-223; radium Ra 223 dichloride; sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sipuleucel-T and radium 223 combination (Experimental): Radium-223 will be administered by intravenous injection over 1 minute at 50kbq (1.35 microcurie) per kg body weight per standard of care every 4 weeks at weeks 0, 4, 8, 12, 16, and 20
  Sipuleucel-T will be administered intravenously per standard of care every 2 weeks at weeks 6, 8, and 10
  Interventions: Drug: Radium-223; Biological: Sipuleucel-T
- sipuleucel-T alone (Active Comparator): Sipuleucel-T will be administered intravenously per standard of care every 2 weeks at weeks 6, 8, and 10
  Interventions: Biological: Sipuleucel-T

INTERVENTIONS:
Drug: Radium-223 — 6 infusions of radium-223 with 3 infusions of sipuleucel-T starting after second dose of radium-223
  Other Names: Xofigo, BAY88-8223
  Arms: sipuleucel-T and radium 223 combination
Biological: Sipuleucel-T — 3 infusions of sipuleucel-T alone
  Other Names: Provenge

SUMMARY:
This clinical trial studies the effect of radium-223 when added to sipuleucel-T for treating castrate-resistant prostate cancer that has spread to the bone. Sipuleucel-T is an autologous cellular immunotherapy designed to stimulate an immune response against prostate cancer. It has been suggested that the immune response may be strengthened by radiation therapy. Therefore this study is testing whether radium-223 added to sipuleucel-T increases the immune response and anti-tumor effect against prostate cancer.

DETAILED DESCRIPTION:
This is a randomized study designed to assess the antigen-specific immune response of sipuleucel-T with or without radium-223. Eligible subjects will be registered and randomly assigned in a 1:1 ratio to receive sipuleucel-T and radium-223 or sipuleucel-T alone.

Subjects in both arms (sipuleucel-T and radium) will undergo a standard 1.5 to 2.0 blood volume leukapheresis, followed approximately 3 days later by an IV infusion of sipuleucel-T. This process will occur a total of 3 times at approximately 2-week intervals. Subjects in Arm 1 will receive a total of 6 infusions of radium-223 at IV dose of 50 kBq/kg at 4-week interval.

All participants are allowed to receive the best supportive care which includes secondary hormonal manipulation as required. No chemotherapy, external-beam radiation, or other radionuclides are allowed while on active treatment but are permitted after completion of active treatment. Glucocorticoid-containing treatments should be minimized to less than the equivalent dose of prednisone 10mg daily if feasible for the 3 months following sipuleucel-T therapy. All patients continue medical or surgical castration during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided prior to initiation of study procedures
2. Age ≥ 18 years
3. Histologically documented adenocarcinoma prostate cancer confirmed by a pathology report from prostate biopsy or a radical prostatectomy specimen. If prostatic tumor is of mixed histology, > 50% of the tumor must be adenocarcinoma
4. Bone metastases as manifested by one or more lesions on a bone scan performed within 2 months of screening
5. Castrate-resistant prostate cancer, in the setting of castrate levels of testosterone (≤ 50 ng/dL), defined as current or historical evidence of disease progression concomitant with surgical castration or androgen deprivation therapy (ADT), as demonstrated by two consecutive rises in PSA OR new lesions on bone scan:

   * PSA progression will be defined as 2 rising PSA values compared to a reference value, measured at least 7 days apart and the second value is ≥ 2 ng/mL [1]. It must be documented within 2 months of screening.
   * Appearance of one or more new areas of abnormal uptake on bone scan when compared to imaging studies acquired during castration therapy or against the precastration studies if there was no response. Increased uptake of pre-existing lesions on bone scan does not constitute progression. It must be documented within 4 months of screening
6. Serum PSA ≥ 2.0 ng/mL
7. Screening ECOG perf status ≤ 1
8. Asymptomatic or minimally symptomatic disease (no narcotic analgesic; other analgesics use is allowed)
9. Prior abiraterone and enzalutamide are permitted, but not required
10. Concurrent osteoclast-inhibitory therapies (zoledronic acid, denosumab) are permitted if patients have been on a stable dose for at least 1 month
11. Adequate screening hematologic, renal, and liver function as evidenced by laboratory test results within the following ranges ≤ 28 days prior to registration:

    * Absolute neutrophil count (ANC) ≥ 1.5 x109/L
    * Platelet count ≥ 100 x109/L
    * Hemoglobin ≥ 10.0 g/dL
    * Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
    * Creatinine ≤ 1.5 x ULN
    * Albumin > 25 g/L

Exclusion Criteria:

1. The presence of known lung or liver metastases greater than 1.0 cm in the long axis diameter
2. The presence of lymphadenopathy greater than 3 cm in the short-axis diameter
3. The presence of known brain metastases
4. Spinal cord compression, imminent long bone fracture, or any other condition that, in the opinion of the investigator, is likely to require radiation therapy and/or steroids for pain control during the active phase
5. Previous treatment with chemotherapy for mCRPC (adjuvant chemotherapy is permitted), or chemotherapy for any reason within 2 years prior to registration
6. Intention to receive chemotherapy within 6 months after enrollment in protocol therapy
7. History of radiation therapy, either via external beam or brachytherapy within 28 days prior to registration
8. Systemic radiotherapy with strontium-89, samarium-153, rhenium-186 or rhenium-188 for the treatment of bony metastases within previous 24 weeks
9. Prior history of other cancers (except non-melanoma skin cancers or low-grade low-stage urothelial cancers)
10. Use of prednisone or equivalent systemic corticosteroid within 2 weeks of treatment. Use of inhaled, intranasal, intra-articular, and topical steroids is allowed. Oral or IV steroids to prevent or treat IV contrast reactions are allowed
11. Use of opioid analgesics for cancer-related pain
12. Use of experimental drug within 4 weeks of treatment
13. Uncontrolled medical conditions including diabetes, heart failure, COPD, ulcerative colitis, or Crohn's disease
14. Uncontrolled fecal incontinence
15. Any medical intervention, any other condition, or any other circumstance which, in the opinion of the investigator, could compromise adherence with study requirements or otherwise compromise the study's objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Antonarakis, MD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Tulane Cancer Center, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marshall CH, Fu W, Wang H, Park JC, DeWeese TL, Tran PT, Song DY, King S, Afful M, Hurrelbrink J, Manogue C, Cotogno P, Moldawer NP, Barata PC, Drake CG, Posadas EM, Armstrong AJ, Sartor O, Antonarakis ES. Randomized Phase II Trial of Sipuleucel-T with or without Radium-223 in Men with Bone-metastatic Castration-resistant Prostate Cancer. Clin Cancer Res. 2021 Mar 15;27(6):1623-1630. doi: 10.1158/1078-0432.CCR-20-4476. Epub 2021 Jan 15. PMID 33451978
- [Derived] Gongora ABL, Marshall CH, Velho PI, Lopes CDH, Marin JF, Camargo AA, Bastos DA, Antonarakis ES. Extreme Responses to a Combination of DNA-Damaging Therapy and Immunotherapy in CDK12-Altered Metastatic Castration-Resistant Prostate Cancer: A Potential Therapeutic Vulnerability. Clin Genitourin Cancer. 2022 Apr;20(2):183-188. doi: 10.1016/j.clgc.2021.11.015. Epub 2021 Dec 24. No abstract available. PMID 35027313

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One screen failure and one withdrew consent prior to randomization, two participants withdrew prior to receiving treatment
Groups:
- Sipuleucel-T and Radium 223 Combination: Radium-223 will be administered by intravenous injection over 1 minute at 50kbq (1.35 microcurie) per kg body weight per standard of care every 4 weeks at weeks 0, 4, 8, 12, 16, and 20
  Sipuleucel-T will be administered intravenously per standard of care every 2 weeks at weeks 6, 8, and 10
  Radium-223: 6 infusions of radium-223 with 3 infusions of sipuleucel-T starting after second dose of radium-223
  Sipuleucel-T: 3 infusions of sipuleucel-T alone
Period: Overall Study
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 6
  >=65 years | 15 | 11 | 26
Age, Continuous [Mean (Full Range); unit: years] | 71.6 [64 to 88] | 70.3 [57 to 86] | 71 [57 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 11 | 10 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Immune Responses to Treatment With Sipuleucel-T (With or Without Radium-223) Measured by Peripheral PA2024 T-cell Proliferation
Description: Peripheral PA2024-specific T-cell proliferation responses using a 3H-thymidine incorporation assay at 6 weeks after the first dose of sipuleucel-T, measured by SI (Stimulation Index [3H-thymidine incorporation in the presence of antigen divided by 3H-thymidine incorporation with media alone] ).
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 16 | 16
fold change | 7.0 [4.12 to 20.2] | 22.4 [17.2 to 31.4]

2. Secondary Outcome: Peripheral PA2024 Specific T-cell Proliferation as Measured by Stimulation Index Over Time
Description: Mean peripheral PA2024 specific T-cell proliferation using a 3H-thymidine incorporation assay reported as SI (Stimulation Index [3H-thymidine incorporation in the presence of antigen divided by 3H-thymidine incorporation with media alone] ) at baseline and 6, 10, 14, 26, 39, and 52 weeks after the first infusion of sipuleucel-T.
Time Frame: Up to 52 weeks
Population: Data was only collected from 13 out of 16 participants in the Sipuleucel-T and radium 223 combination arm and 10 out of 16 participants in the Sipuleucel-T arm
Measure: Mean (Inter-Quartile Range); unit: Stimulation Index
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 13 | 10
Stimulation Index
  Baseline: number analyzed (Participants) | 12 | 10
  Baseline | 1.7 [1.0 to 2.2] | 1.4 [1.2 to 1.5]
  Week 6: number analyzed (Participants) | 12 | 10
  Week 6 | 25.7 [4.4 to 37.0] | 49.8 [30.5 to 44.5]
  Week 10: number analyzed (Participants) | 13 | 8
  Week 10 | 27.8 [8.6 to 34.2] | 42.0 [26.3 to 56.0]
  Week 14: number analyzed (Participants) | 11 | 9
  Week 14 | 23.0 [7.0 to 21.8] | 42.2 [32.1 to 56.1]
  Week 26: number analyzed (Participants) | 9 | 3
  Week 26 | 27.2 [12.2 to 26.4] | 25.6 [15.4 to 36.6]
  Week 39: number analyzed (Participants) | 6 | 1
  Week 39 | 20.7 [5.4 to 22.3] | 25.3 [25.3 to 25.3]
  Week 52: number analyzed (Participants) | 3 | 1
  Week 52 | 16.5 [4.4 to 23.3] | 11.8 [11.8 to 11.8]

3. Secondary Outcome: Time to Radiographic or Clinical Progression
Description: Number of weeks from baseline until radiographic or clinical progression, whichever comes first. Radiographic progression is assessed by RECIST (Response Evaluation Criteria in Solid Tumors) and PCWG2 criteria (Prostate Cancer Working Group 2). Per RECIST, progression is defined as ≥ 20% and ≥ 5 mm from nadir of the sum of the diameters of target lesions. Per PCWG2 criteria, radiographic progression is defined as ≥ 20% sum of the longest diameter of target lesions, or ≥ 2 new lesions on bone scan from baseline. Clinical progression is defined as new spinal cord or nerve root compression, new pathologic fracture or use of opioid analgesics for cancer-related pain.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: WEEKS
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 16 | 16
WEEKS | 38.7 [18.9 to NA] — Upper bound of median not reached, therefore cannot be calculated | 11.9 [8.0 to 15.0]

4. Secondary Outcome: PSA50 Response (at Least a 50% Decline in PSA)
Description: Number of participants with PSA50 response defined as at least a 50% decline in Prostate Specific Antigen (PSA) from baseline value
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 14 | 15
Participants | 0 | 5

5. Secondary Outcome: Peripheral PAP Specific T-cell Proliferation as Measured by Stimulation Index Over Time
Description: Mean peripheral PAP specific T-cell proliferation using a 3H-thymidine incorporation assay reported as SI (Stimulation Index [3H-thymidine incorporation in the presence of antigen divided by 3H-thymidine incorporation with media alone] ) at baseline and 6, 10, 14, 26, 39, and 52 weeks after the first infusion of sipuleucel-T
Time Frame: Up to 52 weeks
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: Stimulation Index
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 13 | 10
Stimulation Index
  Baseline: number analyzed (Participants) | 12 | 10
  Baseline | 1.1 [0.7 to 1.0] | 1.2 [1.0 to 1.4]
  Week 6: number analyzed (Participants) | 12 | 10
  Week 6 | 1.6 [0.9 to 1.4] | 12.5 [1.3 to 4.6]
  Week 10: number analyzed (Participants) | 13 | 8
  Week 10 | 3.1 [0.8 to 3.8] | 5.7 [1.2 to 4.2]
  Week 14: number analyzed (Participants) | 11 | 9
  Week 14 | 2.3 [0.7 to 2.3] | 6.1 [1.0 to 7.9]
  Week 26: number analyzed (Participants) | 9 | 3
  Week 26 | 3.9 [0.7 to 3.8] | 1.5 [1.0 to 1.7]
  Week 39: number analyzed (Participants) | 6 | 1
  Week 39 | 4.1 [1.3 to 3.5] | 1.8 [1.8 to 1.8]
  Week 52: number analyzed (Participants) | 3 | 1
  Week 52 | 2.2 [0.5 to 3.1] | 1.9 [1.9 to 1.9]

6. Secondary Outcome: Peripheral PA2024 Specific T-cell Activation
Description: Mean peripheral PA2024 specific T-cell activation to sipuleucel-T using interferon gamma (IFNγ) enzyme-linked immunosorbent spot (ELISPOT), as measured by cells per 300,000 PBMCs at baseline and weeks 6, 10, 14, 26, 39, and 52 weeks after the first infusion of sipuleucel-T.
Time Frame: Up to 52 weeks
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: cells per 300,000 PBMCs
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 13 | 10
cells per 300,000 PBMCs
  Baseline: number analyzed (Participants) | 12 | 10
  Baseline | 3.6 [1.0 to 1.8] | 6.0 [1.0 to 4.8]
  Week 6: number analyzed (Participants) | 12 | 10
  Week 6 | 66.5 [17.5 to 127.7] | 194.3 [34.2 to 349.8]
  Week 10: number analyzed (Participants) | 13 | 8
  Week 10 | 72.9 [8.0 to 133.7] | 116.4 [14.3 to 232.8]
  Week 14: number analyzed (Participants) | 11 | 9
  Week 14 | 73.6 [17.3 to 115.3] | 137.8 [41.7 to 164.0]
  Week 26: number analyzed (Participants) | 9 | 3
  Week 26 | 87.7 [12.7 to 137.0] | 169.9 [112.7 to 247.8]
  Week 39: number analyzed (Participants) | 6 | 1
  Week 39 | 27.3 [6.4 to 43.8] | 19.0 [19.0 to 19.0]
  Week 52: number analyzed (Participants) | 3 | 1
  Week 52 | 22.4 [12.0 to 33.2] | 26.0 [26.0 to 26.0]

7. Secondary Outcome: Peripheral PAP Specific T-cell Activation
Description: Mean peripheral PAP specific T-cell activation to sipuleucel-T using interferon gamma (IFNγ) enzyme-linked immunosorbent spot (ELISPOT) measured as cells per 300,000 PBMCs at baseline and weeks 6, 10, 14, 26, 39, and 52 weeks after the first infusion of sipuleucel-T.
Time Frame: Up to 52 weeks
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: cells per 300,000 PBMCs
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 13 | 10
cells per 300,000 PBMCs
  Baseline: number analyzed (Participants) | 12 | 10
  Baseline | 0.9 [0.0 to 1.8] | 4.8 [0.0 to 1.7]
  Week 6: number analyzed (Participants) | 12 | 10
  Week 6 | 7.8 [0.0 to 2.8] | 10.9 [0.0 to 18.7]
  Week 10: number analyzed (Participants) | 13 | 8
  Week 10 | 14.1 [0.0 to 3.7] | 19.4 [0.0 to 6.5]
  Week 14: number analyzed (Participants) | 11 | 9
  Week 14 | 12.2 [0.2 to 5.3] | 9.0 [0.0 to 5.0]
  Week 26: number analyzed (Participants) | 9 | 3
  Week 26 | 10.4 [0.7 to 2.3] | 1.0 [0.0 to 1.5]
  Week 39: number analyzed (Participants) | 6 | 1
  Week 39 | 5.0 [0.3 to 2.8] | 1.3 [1.3 to 1.3]
  Week 52: number analyzed (Participants) | 3 | 1
  Week 52 | 3.0 [0.8 to 4.5] | 0.0 [0.0 to 0.0]

8. Secondary Outcome: PA2024 Specific Antibody (IgM) Response
Description: Mean titer of PA2024 specific antibody (IgM) response to sipuleucel-T using enzyme-linked immunosorbent assay (ELISA) at baseline and weeks 6, 10, 14, 26, 39, and 52 weeks after the first infusion of sipuleucel-T.
Time Frame: Up to 52 weeks
Population: Data was only collected from 14 out of 16 participants in the Sipuleucel-T and radium 223 combination arm and 14 out of 16 participants in the Sipuleucel-T arm
Measure: Mean (Inter-Quartile Range); unit: titer
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 14 | 14
titer
  Baseline | 1567.9 [200 to 1600] | 2253.6 [350 to 3200]
  Week 6: number analyzed (Participants) | 12 | 14
  Week 6 | 108941.7 [19400 to 204800] | 164114.3 [102400 to 204800]
  Week 10: number analyzed (Participants) | 13 | 11
  Week 10 | 165434.6 [25600 to 204800] | 214690.9 [128000 to 307200]
  Week 14: number analyzed (Participants) | 11 | 9
  Week 14 | 101422.7 [7200 to 153600] | 185600.0 [102400 to 204800]
  Week 26: number analyzed (Participants) | 11 | 2
  Week 26 | 56586.4 [16000 to 76800] | 28800.0 [17600 to 40000]
  Week 39: number analyzed (Participants) | 9 | 1
  Week 39 | 37338.9 [3200 to 51200] | 204800.0 [204800 to 204800]
  Week 52: number analyzed (Participants) | 4 | 0
  Week 52 | 28400.0 [2800 to 30400] |

9. Secondary Outcome: PA2024 Specific Antibody (IgG) Response
Description: Mean titer of PA2024 specific antibody (IgG) response to sipuleucel-T using enzyme-linked immunosorbent assay (ELISA) at baseline and weeks 6, 10, 14, 26, 39, and 52 weeks after the first infusion of sipuleucel-T.
Time Frame: Up to 52 weeks
Population: as for outcome 8
Measure: Mean (Inter-Quartile Range); unit: titer
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 14 | 14
titer
  Baseline | 382.1 [50.0 to 350] | 771.4 [62.5 to 800]
  Week 6: number analyzed (Participants) | 13 | 14
  Week 6 | 1476.9 [200.0 to 1600] | 7878.6 [1000.0 to 5600]
  Week 10: number analyzed (Participants) | 14 | 11
  Week 10 | 3442.9 [400.0 to 6400] | 23272.7 [1600.0 to 6400]
  Week 14: number analyzed (Participants) | 12 | 9
  Week 14 | 4191.7 [350.0 to 4000] | 15733.3 [800.0 to 3200]
  Week 26: number analyzed (Participants) | 11 | 2
  Week 26 | 3568.2 [1000.0 to 6400] | 7200.0 [4400.0 to 10000]
  Week 39: number analyzed (Participants) | 9 | 1
  Week 39 | 2738.9 [400.0 to 1600] | 25600.0 [25600.0 to 25600]
  Week 52: number analyzed (Participants) | 4 | 0
  Week 52 | 3812.5 [612.5 to 4400] |

10. Secondary Outcome: PAP Specific Antibody (IgG) Response Over Time
Description: Mean titer of PAP specific antibody (IgG) response to sipuleucel-T using enzyme-linked immunosorbent assay (ELISA) at baseline and weeks 6, 10, 14, 26, 39, and 52 weeks after the first infusion of sipuleucel-T.
Time Frame: Up to 52 weeks
Population: as for outcome 8
Measure: Mean (Inter-Quartile Range); unit: titer
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 14 | 14
titer
  Baseline | 796.4 [50 to 800] | 1475.0 [125 to 800]
  Week 6: number analyzed (Participants) | 13 | 14
  Week 6 | 3765.4 [400 to 1600] | 10546.4 [800 to 5600]
  Week 10: number analyzed (Participants) | 14 | 11
  Week 10 | 15125.0 [800 to 11200] | 44563.6 [4800 to 25600]
  Week 14: number analyzed (Participants) | 12 | 8
  Week 14 | 6554.2 [625 to 6400] | 6450.0 [2450 to 12800]
  Week 26: number analyzed (Participants) | 11 | 2
  Week 26 | 5354.5 [400 to 4800] | 51400.0 [25900 to 76900]
  Week 39: number analyzed (Participants) | 9 | 1
  Week 39 | 3916.7 [400 to 6400] | 204800.0 [204800 to 204800]
  Week 52: number analyzed (Participants) | 4 | 0
  Week 52 | 5100 [700 to 8000] |

11. Secondary Outcome: PAP Specific Antibody (IgM) Response
Description: Mean titer of PAP specific antibody (IgM) response to sipuleucel-T using enzyme-linked immunosorbent assay (ELISA) at baseline and weeks 6, 10, 14, 26, 39, and 52 weeks after the first infusion of sipuleucel-T.
Time Frame: Up to 52 weeks
Population: as for outcome 8
Measure: Mean (Inter-Quartile Range); unit: titer
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 14 | 14
titer
  Baseline: number analyzed (Participants) | 14 | 13
  Baseline | 4714.3 [250 to 1600] | 6253.8 [400 to 3200]
  Week 6: number analyzed (Participants) | 11 | 14
  Week 6 | 99209.1 [19200 to 51200] | 112114.3 [16000 to 204800]
  Week 10: number analyzed (Participants) | 13 | 11
  Week 10 | 183184.6 [25600 to 409600] | 210909.1 [76800 to 409600]
  Week 14: number analyzed (Participants) | 12 | 8
  Week 14 | 73250.0 [5200 to 64000] | 238400.0 [166400 to 409600]
  Week 26: number analyzed (Participants) | 11 | 2
  Week 26 | 72363.6 [12800 to 38400] | 205600.0 [103600 to 307600]
  Week 39: number analyzed (Participants) | 8 | 1
  Week 39 | 36425.0 [5600 to 25600] | 409600.0 [409600 to 409600]
  Week 52: number analyzed (Participants) | 4 | 0
  Week 52 | 33200.0 [2800 to 44800] |

12. Secondary Outcome: Sipuleucel-T Product Immune Parameters as Assessed by Number of CD54+ Cells
Description: Mean number of CD54 + cells
Time Frame: Up to 4 weeks
Population: as for outcome 8
Measure: Mean (Inter-Quartile Range); unit: cells x 10 ^ 6
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 14 | 14
cells x 10 ^ 6 | 2730.3 [1704.8 to 3474.5] | 2059.1 [1598.2 to 2512.5]

13. Secondary Outcome: Sipuleucel-T Product Immune Parameters as Assessed by CD54+ Upregulation
Description: Mean CD54+ Upregulation of Sipuleucel-T
Time Frame: Up to 4 weeks
Population: as for outcome 8
Measure: Mean (Inter-Quartile Range); unit: cells x 10^6
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 14 | 14
cells x 10^6 | 29.8 [26.4 to 35.1] | 31.3 [25.1 to 35.1]

14. Secondary Outcome: Sipuleucel-T Product Immune Parameters as Assessed by Total Nucleated Cell Count
Description: Mean number of Total Nucleated Cells
Time Frame: Up to 4 weeks
Population: as for outcome 8
Measure: Mean (Inter-Quartile Range); unit: cells 10^6
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
Number analyzed (Participants) | 14 | 14
cells 10^6 | 11580.5 [7445.2 to 13961.0] | 12740.5 [9127.8 to 14740.2]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sipuleucel-T and Radium 223 Combination | Sipuleucel-T Alone
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/16 | 1/16
Other Adverse Events (participants affected / at risk) | 12/16 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T and Radium 223 Combination (N=16) | Sipuleucel-T Alone (N=16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T and Radium 223 Combination (N=16) | Sipuleucel-T Alone (N=16)
Pain (General disorders) | 12 (12) | 12 (12)
Chills (General disorders) | 2 (2) | 6 (6)
Fatigue (General disorders) | 5 (5) | 3 (3)
Flu Like Symptoms (General disorders) | 4 (4) | 3 (3)
Fever (General disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
White Blood Cell Decreased (Investigations) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 6 (6)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Edema Limbs (General disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Catheter Related Infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT02463799/Prot_SAP_000.pdf